CLINICAL TRIAL: NCT01190241
Title: Targeted Therapy Selection Based on Tumor Tissue Kinase Activity Profiles for Patients With Advanced Solid Malignancies, an Exploratory Study
Acronym: TSAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: VitrOmics BV (Unknown)
Responsible Party: Principal Investigator, M. Labots, medical oncologist, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/124
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Advanced Solid Tumors; Inoperable; Metastasis
Keywords: targeted therapy; individualized medicine; tyrosine kinase inhibitor; kinome profiling; Metastasized
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Sunitinib; Erlotinib Hydrochloride; Everolimus; Lapatinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Targeted treatment (Experimental): Targeted treatment with desatinib or sunitinib or erlotinib or everolimus or lapatinib or sorafenib
  Interventions: Drug: desatinib or sunitinib or erlotinib or everolimus or lapatinib or sorafenib

INTERVENTIONS:
Drug: desatinib or sunitinib or erlotinib or everolimus or lapatinib or sorafenib — The drug will be selected based on ex vivo test on the tumor tissue. The patients will be treated with the selected drug until disease progression.

SUMMARY:
The purpose of this study is to select targeted treatment based on ex vivo kinase activity inhibition profiles to targeted agents of tumor tissue from patients with advanced cancer for whom no standard treatment is available.

DETAILED DESCRIPTION:
Specific signalling proteins that are important for tumor growth can be targeted by agents. These are called targeted agents or targeted treatment. Thus far, it is unclear which patients will respond to these targeted agents. It is assumed that responses to these agents depend on specific receptor and protein signalling activities in tumor tissues. The investigators propose that kinase activity profiling may be a potential clinical diagnostic tool to predict tumor response to targeted treatment with tyrosine kinase inhibitors.

The investigators will determine ex vivo kinase activity inhibition profiles of tumor tissue to different targeted agents. Tumor tissue from patients with advanced cancer for whom no standard treatment is available will be used.

Patients will be treated with the selected targeted agent and the clinical benefit will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with an advanced (unresectable and/or metastatic) solid malignancy for whom no standard treatment is available.
* Patients should have received at least one prior standard medical treatment regimen for their advanced disease.
* Patients with progressive disease within 12 weeks prior to the start of study medication based on radiological assessment.
* At least one tumor lesion should be assessable for biopsy to perform kinase activity analysis.
* Age ≥ 18 years.
* Histological or cytological documentation of cancer is required.
* Patients with at least one measurable lesion. Lesions must be evaluated by CT-scan or MRI according to Response Evaluation Criteria in Solid Tumors (RECIST).
* WHO performance status 0 - 2
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * Hemoglobin ≥ 5.6 mmol/L
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelet count ≥ 100x10*9/l
  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) 22 of 59
  * ALT and AST ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
  * Serum creatinine ≤ 1.5 x ULN or a calculated creatinine clearance ¡Ý 50 ml/min
  * Activated partial thromboplastin time < 1.25 x ULN
  * Prothrombin time or INR < 1.25 x ULN
* Patients should be able to swallow oral medication.
* Written informed consent

Exclusion Criteria:

* History of cardiac disease:

  * Congestive heart failure >NYHA class 2.
  * Active Coronary Artery Disease (myocardial infarction more than 6 months prior to screening is allowed).
  * Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Uncontrolled hypertension. Blood pressure must be ≤ 160/95 mmHg at the time of screening on a stable antihypertensive regimen. Blood pressure must be stable on at least 3 separate measurements on at least 2 separate days.
* Uncontrolled infections (> grade 2 NCI-CTC version 3.0).
* Subjects with serious non-healing wound, ulcer, or bone fracture.
* History or clinical evidence of central nervous system (CNS) disease, including primary brain tumor and brain metastases.
* Clinical findings associated, in the judgment of the investigator, with an unacceptably high tumor biopsy risk
* Pregnant or breast-feeding subjects.
* Concurrent anticancer chemotherapy, immunotherapy or investigational drug therapy during the study or within 4 weeks of the start of study drug.
* Radiotherapy on target lesions during study or within 4 weeks of the start of study drug. Palliative radiotherapy will be allowed.
* Concomitant use of dexamethasone, anti-convulsants and anti-arrhythmic drugs other than digoxin or beta blockers.
* Major surgery within 28 days of start of treatment. The surgical wound should be fully healed prior to the start of study drug. In subjects who experienced wound healing complications during therapy, treatment should be withheld until the wound is fully healed.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject¡-s participation in the study or evaluation of the study results.
* Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The clinical benefit rate (CBR) of this therapy selection approach. | 12 weeks
  The clinical benefit rate (CBR) is defined by the number of patients demonstrating either a complete or partial response or stable disease after 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Henk Verheul, M.D., PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (2):
- Netherlands (2):
  - Medical Center Alkmaar, Alkmaar
  - VU University Medical Center, Amsterdam

REFERENCES:
- [Derived] Labots M, Van der Mijn JC, Dekker H, Ruijter R, Pham TV, Van der Vliet HJ, Van der Hoeven JJM, Meijer GA, Verheul HMW. Selection of Protein Kinase Inhibitors Based on Tumor Tissue Kinase Activity Profiles in Patients with Refractory Solid Malignancies: An Interventional Molecular Profiling Study. Oncologist. 2018 Oct;23(10):1135-e118. doi: 10.1634/theoncologist.2018-0263. Epub 2018 Jul 17. PMID 30018133